CLINICAL TRIAL: NCT01425385
Title: Non-Invasive Assessment of Cerebral Blood Flow Autoregulation in Patients Undergoing Liver Transplantation
Brief Title: Autoregulation Assessment During Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00051645
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Liver Failure; Liver Transplantation; Encephalopathy
Keywords: liver failure; liver transplantation
MeSH Terms: conditions — Liver Failure; Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Autoregulation monitoring: Patients will be grouped into Meld Score
  Interventions: Other: Near infrared spectroscopy monitoring; Other: Autoregulation monitoring

INTERVENTIONS:
Other: Near infrared spectroscopy monitoring — This is an observational study without interventions
  Other Names: Cerebral oximetry index and hemaglobin volume index
Other: Autoregulation monitoring — There are no interventions in this observational study
  Other Names: Cerebral oximetry

SUMMARY:
Patients with liver failure undergoing liver transplantation often have clinical or sub-clinical encephalopathy that may lead to increased intracranial pressure. The latter may lead to abnormal regulation of blood flow to the brain (cerebral autoregulation) complicating patient management during and after general anesthesia. The current methods for monitoring for elevated intracranial pressure are invasive and, thus, limited to severe encephalopathy. In this study the investigators will evaluate the potential utility of monitoring cerebral blood flow (CBF) autoregulation non-invasively using near infra-red spectroscopy in patients undergoing liver transplantation.

DETAILED DESCRIPTION:
Hepatic encephalopathy complicating chronic liver failure in patients undergoing liver transplantation increases the risk for adverse outcomes including mortality. Even mild hepatic encephalopathy may not be recognized clinically without specific testing but can be associated with impaired functional status and reduced quality of life before liver transplantation. The changes that can be seen in chronic liver failure, (cerebral edema and increased intracranial pressure) can adversely affect cerebral blood flow autoregulation that may predispose to brain injury during the multiple hemodynamic perturbations that occur during and after liver transplantation. Currently, invasive monitoring with an intracranial "bolt" is the only method to aggressively manage patients with elevated intracranial pressure from acute liver failure and hepatic encephalopathy. The placement of an intracranial pressure catheter in patient with liver failure is associated with a risk of brain hemorrhage due the presence of a coagulopathy. Further, the risk of this type of monitoring outweighs the benefits in the patients with milder or subclinical forms of hepatic encephalopathy. In this pilot study of 20 patients undergoing liver transplantation the investigators will evaluate the feasibility of non-invasive monitoring of CBF autoregulation and assess whether autoregulation is impaired in this group of patients. The investigators hypothesize that cerebral blood flow autoregulation is impaired in patients undergoing liver transplantation based on severity of liver disease. In this situation, improved patient monitoring would allow clinicians to maintain arterial blood pressure above an individual's lower limit of cerebral blood flow autoregulation that might prevent devastating brain injury during and after surgery. Cerebral blood flow autoregulation can be continuously monitored by evaluating the correlation coefficient between cerebral blood flow velocity measured with transcranial Doppler and arterial blood pressure. The investigators have developed a novel method of autoregulation monitoring using near infrared spectroscopy that allows continuous monitoring of autoregulation with the cerebral oximetry index and the hemoglobin volume index(, a moving linear correlation coefficient between cortical tissue oxygen saturation and hemoglobin level with arterial blood pressure, respectively. The latter approach is more practical and would allow widespread autoregulation monitoring in diverse clinical settings. A secondary hypothesis of this study is that near infrared spectroscopy-based monitoring of CBF autoregulation will provide an accurate assessment of the limits of autoregulation compared with the more clinically challenging transcranial Doppler methods .

Specific Aims:

1. To assess whether patients undergoing liver transplantation have impaired cerebral blood flow autoregulation.
2. To evaluate whether non-invasive monitoring of cerebral blood flow autoregulation with cerebral oximetry index and hemoglobin volume index can identify the lower limit of autoregulation within 10 mmHg compared with that measured with transcranial Doppler.

ELIGIBILITY:
Inclusion Criteria:

-Age > 18 years old and undergoing liver transplantation.

Exclusion Criteria:

* Clinical instability as judged by the attending physicians whereby autoregulation monitoring may interfere with clinical care.
* Women of child bearing potential require a negative urine human chorionic gonadotropin (HCG) test to be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this pilot study we will enroll 20 patients undergoing orthotopic liver transplantation at The Johns Hopkins Hospital. Patients will receive standard care during the procedure. Study related procedures are non-invasive and observational. There will be no interventions based on the results of the study data. The study will include only the immediate operative period. The patients will have transcranial Doppler monitoring and near infrared spectroscopy monitoring during surgery beginning before anesthesia induction and continued until the end of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Hogue, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Zheng Y, Villamayor AJ, Merritt W, Pustavoitau A, Latif A, Bhambhani R, Frank S, Gurakar A, Singer A, Cameron A, Stevens RD, Hogue CW. Continuous cerebral blood flow autoregulation monitoring in patients undergoing liver transplantation. Neurocrit Care. 2012 Aug;17(1):77-84. doi: 10.1007/s12028-012-9721-1. PMID 22644887